CLINICAL TRIAL: NCT00673218
Title: The Effect of Xolair on Inhibiting Leukotriene and Cytokine (IL-4 and IL-13) Release From Blood Basophils
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Creighton University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CIGE025AUS22
Record Dates: First submitted 2008-03-30; First posted 2008-05-07 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Allergy
Keywords: IL13; Cytokines; Basophil stimulation
MeSH Terms: conditions — Hypersensitivity | interventions — Sodium Chloride; Omalizumab; rhuMAb-E25

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Saline injection to match active
  Interventions: Drug: Placebo
- Treatment (Experimental): Active treatment with Xolair 150 to 375 mg is administered SC every 2 or 4 weeks
  Interventions: Drug: Xolair

INTERVENTIONS:
Drug: Placebo — Placebo, Q2 or 4 weeks depending on Ige level and weight as appropriate for active treatment.
  Other Names: Saline
  Arms: 1
Drug: Xolair — 150 to 375 mg is administered SC every 2 or 4 weeks
  Other Names: Omalizumab, rhumab-E25
  Arms: Treatment

SUMMARY:
If you are allergic to ragweed, and not taking certain medications, you will be asked to have blood drawn. We will perform experiments on your blood cells.

DETAILED DESCRIPTION:
Adult ragweed allergic subjects will have blood drawn. Basophils will be enriched and stimulated with allergen and controls. Supernatants from these stimulations will be assayed for cytokines and histamine.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19 to 50
* At least 2 year history of ragweed allergic rhinitis
* Positive skin prick tests to ragweed >5 mm wheal diameter
* IgE <700 iU/m

Exclusion Criteria:

* Use of prohibited medications (e.g. antihistamine in past 7 days and topical or oral corticosteroids in past 1 month, beta-agonist or theophylline for 2 days.
* History of immunotherapy in the past 2 years
* Exposure to Omalizumab in the past 2 years
* Clinically significant non-allergic or perennial rhinitis to avoid mediator release due to environmental allergens
* Asthma other than mild intermittent
* Women of childbearing potential who are not on an accepted form of birth control, as well as women who are breastfeeding
* Known sensitivity to study drug Xolair
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Patients with a previous history of cancer
* Use of any other investigational agent in the last 30 days

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Basophil histamine release | After 4 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Townley, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States